CLINICAL TRIAL: NCT06019728
Title: A Study to Investigate Safety and Tolerability of Higher Infusion Rate to shORten the duraTion of FabrazymE Infusion
Brief Title: A Prospective Study to Investigate Safety and Tolerability of Shorter Infusion of Fabrazyme
Acronym: SHORTEN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS17726; U1111-1287-8570 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Results first posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-09

CONDITIONS: Fabry's Disease
MeSH Terms: conditions — Fabry Disease | interventions — agalsidase beta; Acetaminophen; Diphenhydramine; Dexamethasone; montelukast; Loratadine; Cetirizine; fexofenadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- agalsidase beta (Experimental): agalsidase beta 1 mg/kg infusion once every other week
  Interventions: Drug: AGALSIDASE BETA (GZ419828); Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Dexamethasone; Drug: Montelukast; Drug: Loratadine; Drug: Cetirizine; Drug: Fexofenadine

INTERVENTIONS:
Drug: AGALSIDASE BETA (GZ419828) — Pharmaceutical form: Lyophilized powder for reconstitution Route of administration: IV infusion
  Other Names: Fabrazyme
Drug: Acetaminophen — Tablet or solution; Oral
Drug: Diphenhydramine — Tablet or solution; Oral
Drug: Dexamethasone — Tablet or solution; Oral
Drug: Montelukast — Tablet or chewable tablet or oral granules; Oral
Drug: Loratadine — Tablet or chewable tablet; Oral
Drug: Cetirizine — Tablet or oral solution; Oral
Drug: Fexofenadine — Tablet or oral suspension; Oral

SUMMARY:
This Phase 4 study will evaluate the safety and tolerability of Fabrazyme at current approved dose with increases in the infusion rate and reduced infusion volume. This study aims to generate data to provide the guidance on how infusion rate can be safely increased and minimize the burden of the life-long treatment with Fabrazyme.

DETAILED DESCRIPTION:
The total duration will be up to 7 months

ELIGIBILITY:
Inclusion Criteria:

- Participants with confirmed diagnosis of FD who are ≥2 and ≤65 years of age at the time of signing the informed consent form (ICF) or assent, if applicable.

* Cohort 1: female participants with body weight ≥30 kg who have been treated with Fabrazyme for at least 3 months without IARs during the most recent 3 infusions.
* Cohort 2: non-classic male participants with body weight ≥30 kg who have been treated with Fabrazyme for at least 3 months without IARs during the most recent 3 infusions.
* Cohort 3: classic male participants with body weight ≥30 kg who have been treated with Fabrazyme for at least 3 months without IARs during the most recent 3 infusions.
* Cohort 4: participants with body weight <30 kg who have been treated with Fabrazyme for at least 3 months without IARs during the most recent 3 infusions.

Women of childbearing potential must use a highly effective method of contraception through the study.

Exclusion Criteria:

* Female participants who are pregnant or breastfeeding.
* History of significant allergic disease or hypersensitivity to Fabrazyme or other medicinal products.
* Contraindication to Fabrazyme or any of the premedications or rescue medications (diphenhydramine, loratadine, cetirizine, fexofenadine, acetaminophen, montelukast, dexamethasone).
* Any other medical condition considered to make the increased infusion rate not tolerable at the Investigator's discretion.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (5):
- United States (5):
  - UCLA Medical Center Site Number : 1003, Santa Monica, California
  - Emory University School of Medicine Site Number : 1005, Atlanta, Georgia
  - Infusion Associates Site Number : 1001, Grand Rapids, Michigan
  - Metropolitan Hospital Center Site Number : 1004, New York, New York
  - Lysosomal and Rare Disorders Research and Treatment Center, Inc Site Number : 1002, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LPS17726 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25537&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 4 centers in United States. A total of 8 participants were screened from 10 November 2023 to 27 August 2024, of which none were screen failures.
Pre-assignment Details: A total of 8 participants were enrolled in the study. All participants received same dose in this single-group, single arm study as pre-specified in the protocol and statistical analysis plan (SAP). Note: Reason for not completed = Reason for permanent full study treatment discontinuation.
Groups:
- Fabrazyme®: All participants received Fabrazyme® 1 milligram per kilogram (mg/kg) every 2 weeks (Q2W) via intravenous (IV) infusion for up to 16 weeks (up to 9 infusions).
Period: Overall Study
Arm/Group | Fabrazyme®
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) analysis set included all participants who were enrolled and allocated to study treatment.
Groups:
- Fabrazyme®: All participants received Fabrazyme® 1 mg/kg Q2W via IV infusion for up to 16 weeks (up to 9 infusions).
Arm/Group | Fabrazyme®
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (17.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Reduction in Shortest Tolerated Infusion Duration From Pre-study Average of Recent 3 Infusions
Description: Percent reduction was with respect to the shortest tolerated infusion for the participant. The shortest infusion duration tolerated was the actual shortest duration (highest infusion rate) of a completed infusion tolerated by the participant without experiencing a second infusion associated reaction (IAR). The pre-study infusion duration was derived as the average of the duration of 3 most recent infusions the participant received prior to participating to this study. Percent reduction of infusion duration was calculated as: 100 x (average of pre-study infusion duration [minutes] - actual shortest infusion duration tolerated [minutes]) / average of pre-study infusion duration (minutes).
Time Frame: Up to 16 weeks
Population: The ITT analysis set included all participants who were enrolled and allocated to study treatment.
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Fabrazyme®
Number analyzed (Participants) | 8
percent | 84.19 [80.56 to 86.32]

2. Primary Outcome: Shortest Actual Tolerated Infusion Duration
Description: The shortest infusion duration tolerated was the actual shortest duration (highest infusion rate) of a completed infusion tolerated by the participant without experiencing a second IAR. IARs were events recorded as adverse event of special interest (AESI) and were defined as AEs the Investigator considered related to Fabrazyme® infusion, that occurred on same day as infusion and only after infusion had begun.
Time Frame: Up to 16 weeks
Population: The ITT analysis set included all participants who were enrolled and allocated to study treatment.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Fabrazyme®
Number analyzed (Participants) | 8
minutes | 20.00 [20.00 to 20.00]

3. Secondary Outcome: Number of Participants Who Achieved the Shortest Planned Duration of Infusion Time Without Experiencing Any Infusion Associated Reaction
Description: Number of participants who achieved the shortest planned duration of infusion time without experiencing any IAR is reported. ARs were events recorded as AESI and were defined as AEs the Investigator considered related to Fabrazyme® infusion, that occurred on same day as infusion and only after infusion had begun.
Time Frame: Up to 16 weeks
Population: The ITT analysis set included all participants who were enrolled and allocated to study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Fabrazyme®
Number analyzed (Participants) | 8
Participants | 8

4. Secondary Outcome: Number of Participants Who Achieved the Shortest Planned Duration of Infusion Time Without Experiencing a Second Infusion Associated Reaction
Description: Number of participants who achieved the shortest planned duration of infusion time without experiencing a second IAR is reported. ARs were events recorded as AESI and were defined as AEs the Investigator considered related to Fabrazyme® infusion, that occurred on same day as infusion and only after infusion had begun.
Time Frame: Up to 16 weeks
Population: The ITT analysis set included all participants who were enrolled and allocated to study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Fabrazyme®
Number analyzed (Participants) | 8
Participants | 8

5. Secondary Outcome: Number of Participants Who Tolerated Planned Infusion Duration Shorter Than 90 Minutes Without Experiencing Any Infusion Associated Reaction
Description: Number of participants who tolerated the shortest planned duration of infusion time without experiencing any IAR is reported. ARs were events recorded as AESI and were defined as AEs the Investigator considered related to Fabrazyme® infusion, that occurred on same day as infusion and only after infusion had begun. Participants with an initial planned target duration <90 minutes were considered a responder if they tolerated at least 1 infusion during the study treatment period with actual duration <90 minutes.
Time Frame: Up to 16 weeks
Population: The ITT analysis set included all participants who were enrolled and allocated to study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Fabrazyme®
Number analyzed (Participants) | 8
Participants | 8

6. Secondary Outcome: Number of Participants Who Tolerated Planned Infusion Duration Shorter Than 90 Minutes Without Experiencing a Second Infusion Associated Reaction
Description: Number of participants who tolerated the shortest planned duration of infusion time without experiencing a second IAR is reported. ARs were events recorded as AESI and were defined as AEs the Investigator considered related to Fabrazyme® infusion, that occurred on same day as infusion and only after infusion had begun. Participants with an initial planned target duration <90 minutes were considered a responder if they tolerated at least 1 infusion during the study treatment period with actual duration <90 minutes.
Time Frame: Up to 16 weeks
Population: The ITT analysis set included all participants who were enrolled and allocated to study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Fabrazyme®
Number analyzed (Participants) | 8
Participants | 8

7. Secondary Outcome: Number of Participants Who Tolerated Each Planned Infusion Duration Without Experiencing Any Infusion Associated Reaction
Description: Number of participants who tolerated each planned infusion duration without experiencing any IAR is reported. ARs were events recorded as AESI and were defined as AEs the Investigator considered related to Fabrazyme® infusion, that occurred on same day as infusion and only after infusion had begun. The planned duration of infusion time was 120 minutes, 90 minutes, 60 minutes, 40 minutes, and 20 minutes.
Time Frame: Up to 16 weeks
Population: The ITT analysis set included all participants who were enrolled and allocated to study treatment. Only those participants with data collected at specified timepoints are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Fabrazyme®
Number analyzed (Participants) | 8
Participants
  120 minutes: number analyzed (Participants) | 6
  120 minutes | 6
  90 minutes: number analyzed (Participants) | 7
  90 minutes | 7
  60 minutes | 8
  40 minutes | 8
  20 minutes | 8

8. Secondary Outcome: Number of Participants Who Tolerated Each Planned Infusion Duration Without Experiencing a Second Infusion Associated Reaction
Description: Number of participants who tolerated each planned infusion duration without experiencing a second IAR is reported. ARs were events recorded as AESI and were defined as AEs the Investigator considered related to Fabrazyme® infusion, that occurred on same day as infusion and only after infusion had begun. The planned duration of infusion time was 120 minutes, 90 minutes, 60 minutes, 40 minutes, and 20 minutes.
Time Frame: Up to 16 weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Fabrazyme®
Number analyzed (Participants) | 8
Participants
  120 minutes: number analyzed (Participants) | 6
  120 minutes | 6
  90 minutes: number analyzed (Participants) | 7
  90 minutes | 7
  60 minutes | 8
  40 minutes | 8
  20 minutes | 8

ADVERSE EVENTS:
Time Frame: Adverse events and all-cause mortality were collected from the first dose of study treatment (Day 1) up to 16 weeks
Description: Analysis was performed on the safety analysis set which included all participants who received any amount of study drug (Fabrazyme®) during study treatment period.
Arm/Group | Fabrazyme®
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fabrazyme® (N=8)
Influenza (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Globotriaosylsphingosine Increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2024-07-09): https://cdn.clinicaltrials.gov/large-docs/28/NCT06019728/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT06019728/SAP_001.pdf